CLINICAL TRIAL: NCT02372968
Title: Use of Metabonomics and Body Imaging for Metabolic Health Assessment
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 08.03.MET
Record Dates: First submitted 2015-02-04; First posted 2015-02-26 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2015-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Full body composition and of plasma and urine metabolites — Full body composition in lean, fat and bone mass will be assessed from DXA scans.
  Plasma and urine metabolites will be measured using metabolomics

SUMMARY:
The aim of this pilot study is to develop at Nestlé Research Center a database of metabolic profiles, body composition, food habits and physical activities on a large cohort of human volunteers. Analysis of collected data will serve to measure the variability of the data and to assess the potential of combining metabonomics with imaging techniques (iDXA) to monitor the metabolic and physiologic effects of foods.

DETAILED DESCRIPTION:
The study will be carried out at the metabolic unit of the Nestlé Research Center (Lausanne). A large cohort of subjects will be recruited among Nestlé employees. Body composition will be determined by iDXA (Dual-energy X-ray absorptiometry) and basal metabolism will be measured by metabonomic analysis of urine and plasma samples.

Individual food habits and physical activities will be assessed by questionnaires.

The clinical protocol plans also the measurement of energy expenditure (EE) by indirect calorimetry on a subset of twenty subjects. These EE data will be used to validate iDXA outcomes for resting energy expenditure.

The volunteers can participate a second time to this study in the case they would like to control the evolution of their body composition and metabolism after a period of dietary regime or physical training. In such a case, a minimum period of two months between the visits is required.

After two days of dietary restrictions, the volunteers will come in the morning at the metabolic unit at fasting state, for urine and blood sampling. The metabolism of some foods can bias the metabonomic analyses. Therefore, the consumption of alcoholic beverages, fish meals, liquorice, grapefruit, power drinks and bars, spices, mineral supplements, soft drinks, chocolate, coffee and tea limited to 2 cups per day, are not allowed during two days preceding the visit. In addition, the intake of pain-killers or antiinflammatory drugs is forbidden during the two days before the sampling of urine and blood because their metabolism alters the metabolic profiles of blood and urine.

Antibiotics alter gut microflora, for which the activity represents an important contributor to the urinary metabolic profile. In order to preserve gut microflora-related metabolic information, we recommend a minimum period of one month between the end of any antibiotic therapy and the visit at the metabolic unit.

On the visit day, subjects will come fasting at the metabolic unit, where they will have to:

* Answer some medical questions during an interview with the doctor in charge of the study
* Fill in two questionnaires on food habits and physical activities. A dietician of the CHUV will visit you at NRC to ask you for some questions relative to your food habits. This is to validate the new questionnaire you filled in
* Give a sample of urine
* Undergo iDXA scan (2 consecutive measures will be run at each of the two visits, in order to assess the intra-individual variability of the results) and measure of the state of hydration by bioimpedance The analysis of plasma samples is recommended to complete the metabonomic analysis. However, the blood sampling will be freely decided by each participant. The protocol plans also to perform measurements of resting energy expenditure by indirect calorimetry on a subset of twenty subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects must comply with all the following inclusion criteria:

* Having respected dietary restrictions 2 days before the visit
* Having obtained his/her or his/her legal representative's informed consent

Exclusion Criteria:

Subjects representing one or more of the following criteria are excluded from participation in the study:

* Pregnancy as per precaution principal to avoid risks linked to X-ray exposure
* Any pathology (infectious or other) having required an antibiotic therapy within

  1 month prior to the beginning of the study
* Any therapy (contraception apart) within the 2 days before the visit day
* Subject who cannot be expected to comply with measures
* Currently participating or having participated in another clinical trial during the last 3 months prior to the beginning of this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Studied population: 100-300 subjects, men and women selected out of Nestlé employees
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Lean, fat, and bone mass (Measure of full body composition in lean, fat, and bone mass) | change of body composition after a period of 2 months following baseline
  Measure of full body composition in lean, fat, and bone mass
Screening of metabolites in plasma in fasting condition | Change of plasma metabolites after a period of 2 months post baseline
  Measure of plasma metabolites by Nuclear Magnetic Resonance spectroscopy and Mass Spectrometry
Screening of urine metabolites in fasting condition | Change of urine metabolites after a period of 2 months post baseline
  Measure of urine metabolites by Nuclear Magnetic Resonance spectroscopy and Mass Spectrometry
Food habits (Measure of food habits based on Food Frequency Questionnaires) | Change of food habits after a period of 2 months post baseline
  Measure of food habits based on Food Frequency Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Serge Rezzi, PhD, Study Director — Nestlé Institute of Health Sciences

REFERENCES:
- [Derived] Wei R, Ross AB, Su M, Wang J, Guiraud SP, Draper CF, Beaumont M, Jia W, Martin FP. Metabotypes Related to Meat and Vegetable Intake Reflect Microbial, Lipid and Amino Acid Metabolism in Healthy People. Mol Nutr Food Res. 2018 Nov;62(21):e1800583. doi: 10.1002/mnfr.201800583. Epub 2018 Aug 28. PMID 30098305